CLINICAL TRIAL: NCT01512719
Title: POEM a Novel Endoscopic Treatment for Achalasia
Brief Title: POEM- Peroral Endoscopic Myotomy for Esophageal Motility Disorders
Acronym: POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040411-HMO-CTIL
Record Dates: First submitted 2012-01-15; First posted 2012-01-19 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-03

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- POEM procedure (Experimental): Patients with achalasia that undergo POEM
  Interventions: Procedure: POEM

INTERVENTIONS:
Procedure: POEM — Per Oral Endoscopic Myotomy for achalasia

SUMMARY:
POEM has recently described as an alternative treatment for achalasia in humans. In this procedure the esophageal sphincter is incised through a submucosal tunnel in the esophagus. In this study we aim to perform POEM on achalasia patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Achalasia whom are candidates for Heller Myotomy

Exclusion Criteria:

* Perforation of LES during dilatation
* Pregnant women
* mentally ill patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Resolution of dysphagia | up to 6 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Mintz, MD, Principal Investigator — Hadassah Medical Organization
Locations (3):
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Hadassah Medical Organization, Jerusalem
  - Hadassah Medical Organization Ein-Kerem campus, Jerusalem